CLINICAL TRIAL: NCT01246804
Title: The Influence of GINkGo Biloba on the Pharmacokinetics of the UGT Substrate raltEgraviR (GINGER)
Acronym: GINGER
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: UMCN-AKF 10.02
Record Dates: First submitted 2010-11-22; First posted 2010-11-23 (Estimated); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: HIV Infections; Depression; Mild Cognitive Impairment
Keywords: HIV infections; interaction; pharmacokinetics
MeSH Terms: conditions — HIV Infections; Depression; Cognitive Dysfunction | interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ginkgo biloba + raltegravir (Experimental): 15 days ginkgo biloba 120mg BID + raltegravir 400mg SD
  Interventions: Drug: raltegravir single dose; Drug: ginkgo biloba multiple dose
- raltegravir (Active Comparator): single dose raltegravir 400mg
  Interventions: Drug: raltegravir single dose

INTERVENTIONS:
Drug: raltegravir single dose — single dose 400mg raltegravir
  Other Names: Isentress
Drug: ginkgo biloba multiple dose — 15 days ginkgo biloba 120mg BID
  Other Names: Tavonin
  Arms: ginkgo biloba + raltegravir

SUMMARY:
The objective of this study is to evaluate the effect of ginkgo biloba (steady state) on the pharmacokinetics of a single dose of the UGT-substrate raltegravir. Furthermore the safety profile of the combination is studied.

DETAILED DESCRIPTION:
Ginkgo biloba is an alternative medicine that is popular among HIV-infected patients because if its claimed positive effects on memory, concentration and depression. Alternative medicine can cause drug-drug interactions with regular HIV-medication. Raltegravir is a newly developed HIV integrase inhibitor. It is metabolized in the liver by UGT1A1 and therefore its pharmacokinetic profile can be influenced by inhibitors or inducers of UGT1A1. So far there are no data of the potential effect of ginkgo biloba on glucuronidation in vivo. The current study is designed to evaluate the potential inductive effect of ginkgo biloba on the pharmacokinetics of raltegravir and the safety profile when used in combination.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 and not older than 55 years at screening.
* Subject does not smoke more than 10 cigarettes, 2 cigars, or 2 pipes per day for at least 3 months prior to the first dosing
* Subject has a Quetelet Index (Body Mass Index) of 18 to 30 kg/m2, extremes included.
* Subject is able and willing to sign the Informed Consent Form prior to screening evaluations.
* Subject is in good age-appropriate health condition as established by medical history, physical examination, electrocardiography, results of biochemistry, haematology and urinalysis testing within 4 weeks prior to Day 1. Results of biochemistry, haematology and urinalysis testing should be within the laboratory's reference ranges. If laboratory results are not within the reference ranges, the subject is included on condition that the Investigator judges that the deviations are not clinically relevant. This should be clearly recorded.
* Subject has a normal blood pressure and pulse rate, according to the Investigator's judgement.

Exclusion Criteria:

* Documented history of sensitivity/idiosyncrasy to medicinal products or excipients.
* Positive HIV test.
* Positive hepatitis B or C test.
* Pregnant female (as confirmed by an HCG test performed less than 4 weeks before Day 1) or breast-feeding female. Female subjects of childbearing potential without adequate contraception, e.g. hysterectomy, bilateral tubal ligation, (non-hormonal) intrauterine device, total abstinence, double barrier methods, or two years post-menopausal. They must agree to take precautions in order to prevent a pregnancy throughout the entire conduct of the trial.
* Therapy with any drug (for two weeks preceding dosing), except for paracetamol.
* Relevant history or presence of pulmonary disorders (especially COPD), cardiovascular disorders, neurological disorders (especially seizures and migraine), psychiatric disorders, gastro-intestinal disorders, renal and hepatic disorders, hormonal disorders (especially diabetes mellitus), coagulation disorders.
* Relevant history or current condition that might interfere with drug absorption, distribution, metabolism or excretion.
* History of or current abuse of drugs, alcohol or solvents.
* Inability to understand the nature and extent of the trial and the procedures required.
* Participation in a drug trial within 60 days prior to Day 1.
* Donation of blood within 60 days prior to Day 1.
* Febrile illness within 3 days before Day 1.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2010-11; Primary Completion 2011-03 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
raltegravir concentrations | pharmacokinetic curve after a single dose of raltegravir alone or added to steady state ginkgo biloba
  To determine the effect of chronic use of ginkgo biloba on the single-dose pharma-cokinetics (AUC0-inf, AUC0-12, Cmax, C12) of raltegravir 400mg in healthy volunteers.

SECONDARY OUTCOMES:
adverse events | during entire study
  To determine the safety of a single dose of raltegravir 400mg when combined with chronic use of ginkgo biloba.

CONTACTS AND LOCATIONS:
Overall Officials: David M Burger, PharmD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- CRCN, Radboud University Medical Centre, Nijmegen, Netherlands

REFERENCES:
- See also: Publication of results of the study — http://www.ncbi.nlm.nih.gov/pubmed/22802250